CLINICAL TRIAL: NCT02189317
Title: Liposomal Bupivacaine for Pain Control Following Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Xerogeanes, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00073168
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel (Experimental): This arm will receive Exparel
  Interventions: Drug: Exparel
- Control (No Intervention)

INTERVENTIONS:
Drug: Exparel — For the treatment group a total of 40 cc consisting of 20 cc of 1.3% Exparel® and 20 cc of 0.5 % marcaine will be administered to the ACL harvest site, into the periosteum surrounding the distal tibial tunnel site, and in the proximity of the skin incisions. No infiltration of Exparel will be provided intra-articularly.
  Other Names: Liposomal Bupivacaine
  Arms: Exparel

SUMMARY:
This study will consist of 80 patients ages 18 to 50 at the Emory Orthopaedic and Spine Center who are undergoing Anterior Cruciate Ligament (ACL) reconstruction with a quadriceps tendon autograft or bone patellar tendon bone autograft by Dr. Karas or Dr. Xerogeanes. Patients will be randomized into treatment and control arms. The treatment arm will include 40 patients receiving liposomal bupivacaine intra-operatively in addition to the current standard pain control regimen. The control group will include 40 patients receiving the standard post-operative pain control regimen. Patients will be assessed to identify differences in post-operative pain, satisfaction, as well as concomitant pain medication use. Post-operative range of motion will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 50 chronological years undergoing ACL reconstruction using a quadriceps tendon or BTB autograft.

Exclusion Criteria:

* Patients with known allergies to local anesthetics
* pregnant patients
* patients with a history of liver disease
* patients undergoing bilateral procedures
* Patients undergoing revision ACL surgery and patients undergoing ACL reconstruction using pediatric physeal sparing techniques
* Patients will also be excluded if any clinically significant event or condition is discovered during the time of, or after surgery that may render them medically unstable, or subject them to a surgical complication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Xerogeanes, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Orthopaedic and Spine Center, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Premkumar A, Samady H, Slone H, Hash R, Karas S, Xerogeanes J. Liposomal Bupivacaine for Pain Control After Anterior Cruciate Ligament Reconstruction: A Prospective, Double-Blinded, Randomized, Positive-Controlled Trial. Am J Sports Med. 2016 Jul;44(7):1680-6. doi: 10.1177/0363546516640772. Epub 2016 Apr 25. PMID 27159290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an ambulatory surgery center from July 2014 to March 2015.
Pre-assignment Details: Of the fifty participants who consented for the study, 18 participants who had different graph types were excluded to avoid a potential confounder. Thirty two participants were included in the overall study who had identical graph types.
Groups:
- Bupivacaine HCl: Participants undergoing primary anterior cruciate ligament (ACL) reconstruction with a soft tissue quadriceps tendon autograft received a femoral block immediately before surgery. Participants then received 20 mL 0.25% bupivacaine HCl and 20 ml 0.9% injectable saline administered into the graft harvest site and portal sites during surgery.
- Exparel (Bupivacaine Liposome): Participants undergoing primary anterior cruciate ligament (ACL) reconstruction with a soft tissue quadriceps tendon autograft received a femoral block immediately before surgery. Participants then received a 40-mL suspension of 20 mL Exparel (1 vial of bupivacaine liposome injectable suspension) and 20 mL 0.9% injectable saline administered into the graft harvest site and portal sites during surgery.
Period: Overall Study
Arm/Group | Bupivacaine HCl | Exparel (Bupivacaine Liposome)
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exparel (Liposomal Bupivacaine): Participants undergoing primary anterior cruciate ligament (ACL) reconstruction with a soft tissue quadriceps tendon autograft received a femoral block immediately before surgery. Participants then received a 40-mL suspension of 20 mL Exparel (1 vial of bupivacaine liposome injectable suspension) and 20 mL 0.9% injectable saline administered into the graft harvest site and portal sites during surgery.
- Total: Total of all reporting groups
Arm/Group | Bupivacaine HCl | Exparel (Liposomal Bupivacaine) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Numerical Rating Scale (NRS) Pain Score
Description: The numerical rating scale (NRS) pain score is a self-reported pain scale from 0 to 10 where zero is equal to "no pain" and ten is equal to "worst possible" pain. The score was recorded every 12 hours for up to 144 hours (six days) post-operatively.
Time Frame: Day of Surgery, Post-Operative Day 6 (Up to 144 hours)
Population: Participants who underwent ACL reconstruction surgery and returned a completed post-operative pain and medication journal (bupivacaine HCl group).
  Participants who underwent ACL reconstruction surgery, returned a completed post-operative pain and medication journal, and did not require reoperation (Exparel liposomal/bupivacaine group).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine HCl | Exparel (Liposomal Bupivacaine)
Number analyzed (Participants) | 15 | 14
units on a scale
  Baseline (recovery room) | 3.6 (2.1) | 4.7 (2.0)
  Evening on the day of surgery | 5.0 (3.7) | 4.1 (2.3)
  Day 1 Morning | 5.7 (2.5) | 4.5 (2.1)
  Day 1 Evening | 5.2 (2.6) | 5.6 (1.7)
  Day 2 Morning | 5.1 (2.6) | 4.9 (2.5)
  Day 2 Evening | 4.1 (2.4) | 4.7 (1.9)
  Day 3 Morning | 3.7 (2.5) | 4.8 (1.7)
  Day 3 Evening | 3.6 (2.5) | 4.5 (2.0)
  Day 4 Morning | 3.3 (2.2) | 4.1 (2.0)
  Day 4 Evening | 3.0 (2.0) | 3.6 (2.1)
  Day 5 Morning | 3.3 (2.1) | 2.8 (2.5)
  Day 5 Evening | 3.1 (2.1) | 2.5 (2.4)
  Day 6 Morning | 3.3 (2.2) | 2.5 (2.4)
  Day 6 Evening | 2.4 (2.3) | 1.4 (2.2)

2. Secondary Outcome: Change in Home Opioid Use
Description: The difference in amount of Percocet (7.5/325 tablets) usage post-surgery.
Time Frame: Day of Surgery, Post-Operative Day 6 (Up to 144 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: miligrams
Arm/Group | Bupivacaine HCl | Exparel (Liposomal Bupivacaine)
Number analyzed (Participants) | 15 | 14
miligrams
  Up to 72 hours | 10.2 (4.8) | 9.3 (6.9)
  Day of Surgery | 1.6 (1.3) | 2.5 (1.5)
  Postoperative Day 1 | 4.9 (2.9) | 4.1 (3.2)
  Postoperative Day 2 | 4.0 (2.1) | 2.3 (2.5)
  Postoperative Day 3 | 2.3 (1.9) | 1.3 (1.5)
  Postoperative Day 4 | 1.7 (1.4) | 0.8 (1.0)
  Postoperative Day 5 | 1.6 (1.5) | 0.2 (0.4)
  Postoperative Day 6 | 1.6 (1.6) | 0.3 (0.5)

3. Secondary Outcome: Difference in Time to First Opioid Use
Description: The time difference in hours to first Percocet (7.5/325 tablets) usage post-surgery.
Time Frame: Day of Surgery, Post-Operative Day 6 (Up to 144 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bupivacaine HCl | Exparel (Liposomal Bupivacaine)
Number analyzed (Participants) | 15 | 14
hours | 3.2 (2.1) | 3.1 (0.7)

ADVERSE EVENTS:
Arm/Group | Bupivacaine HCl | Exparel (Bupivacaine Liposome)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine HCl (N=16) | Exparel (Bupivacaine Liposome) (N=16)
Post-operative Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study lacked a third comparison group of participants who received placebo which may have provided another internal control. Additionally, there was a difference in the total milligrams of bupivacaine administered in each study group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes